CLINICAL TRIAL: NCT03462888
Title: Clinico-biological Study/Characterization of Rhabdomyosarcoma in AYA (Adolescents and Young Adults, 15-25-year-old Patients)
Brief Title: Clinico-biological Study/Characterization of Rhabdomyosarcoma in Adolescents and Young Adults, 15-25-year-old Patients
Acronym: RMS-AJA-1701
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Centre Leon Berard (Other); Société Française de lutte contre les Cancers et les leucémies de l'Enfant et l'adolescent (Unknown); French Sarcoma Group (Other); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: RMS-AJA-1701
Record Dates: First submitted 2018-02-26; First posted 2018-03-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Rhabdomyosarcoma
Keywords: Rhabdomyosarcoma; Adolescents and young adults; prognostic factors; molecular profiling
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue extracted at diagnosis from biopsy or from surgical resection of the primary tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rhabdomyosarcoma (RMS) stands for the most frequent soft tissue sarcoma in children and, adolescents and young adults (AYA, 15-25-year-old population), accounting for approximately half of the whole soft tissue sarcomas in these populations.. Conversely, RMS represents a very small proportion of the soft tissue sarcomas in adults (3%), that is less than 1% of all solid cancers of adults.

To date, previous studies undertaken among the paediatric population have pointed out several prognostic factors such as tumor localisation, tumor invasiveness at diagnosis, tumor size, histological subset, and treatment plans. Age at diagnosis remains an independent prognostic factor.

RMS management is consensual in Europe for paediatric population, essentially based on the protocol RMS 2005 within the framework of the European Paediatric Soft tissue sarcoma Study Group (EpSSG). Care in AYAs remain heterogeneous and are either achieved in paediatric department, according to EpSSG guidelines, or in oncology department, known as "adult unit", depending on ESMO (European Society for Medical Oncology), which are non-specific recommendations for the management of rhabdomyosarcoma.

No consensus has been published yet for RMS in AYA despite the growing interest in cancers in AYA population - topic.supported by the French National Cancer Institute (INCa) - and the increasing network between paediatricians and adult-oncologists. Thus management of RMS in AYA remains patchy/unequal depending on the type of care unit.

Herein, with the support of the Oscar Lambret Center, we aim at assessing and identifying clinico-biological prognostic factors of rhabdomyosarcoma in AYA. Eventually, we hope to offer a standardized treatment to this population. Data collected from medical file will be anonymised in a confidential database of which the recipient is the sponsor of the study.

The ancillary study will aim at characterizing the molecular profile of the difficult-to-classify RMS subtypes (fusiform or pleomorphic subsets) in molecular biology for ambiguous cases.

From a scientific point of view, this study aims at understanding the parameters that may influence the prognosis of RMS in AYAs by evaluating various clinical and biological factors.

Biologically, molecular profiling of RMS in AYA may improve the characterization of this tumour in this age group.

At the clinical level, the completeness of the data collected will lead to a better description of RMS in AYAs. We hope to harmonize their therapeutic management by providing therapeutic adjustments according to population subsets.

Finally, these results could also help to adapt the therapeutic management of AYAs within the framework of the European protocol that is currently under construction, and will involve both children and adults.

DETAILED DESCRIPTION:
Rhabdomyosarcoma (RMS) is a rare tumor, with an incidence rate estimated at 4.5-6.9/1,000,000 in paediatric and, adolescent and young adult (AYA, 15 -25 years old) populations. RMS stands for the most frequent soft tissue sarcoma in children and adolescents, accounting for approximately half of the whole soft tissue sarcomas in these populations. Conversely, RMS represents a very small proportion of the soft tissue sarcomas in adults (3%), that is less than 1% of the solid cancers of the adult. To date, previous studies undertaken among the paediatric population have pointed out several prognostic factors such as tumor localisation, tumor invasiveness at diagnosis, tumor size, histological subset, and treatment plans. Age at diagnosis remains an independent prognostic factor. MYOD1 gene expression profile, more common in AYA, also seems to impair the prognosis.

RMS management is consensual in Europe for paediatric population, essentially based on the protocol RMS 2005 within the framework of the European Paediatric Soft tissue sarcoma Study Group (EpSSG). Care in AYAs remain heterogeneous and are either achieved in paediatric department, according to EpSSG guidelines, or in oncology department, known as "adult unit", depending on ESMO (European Society for Medical Oncology), which are non-specific recommendations for the management of rhabdomyosarcoma.

No consensus has been published yet for RMS in AYA despite the growing interest in cancers in AYA population - topic.supported by the French National Cancer Institute (INCa) - and the increasing network between paediatricians and adult-oncologists. Thus management of RMS in AYA remains patchy/unequal depending on the type of care unit.

Principal study

* To evaluate the prognostic value in terms of Progression Free Survival (PFS), in AYA patients with RMS, of clinical factors known as prognostic in children, and of biological factors (MYOD1 mutation in non-alveolar tumor; FOXO1).
* To describe clinical, histological and biological characteristics of RMS in AYA.
* To describe the therapeutic strategy according to the type of department (pediatric, AYA or adults):
* To evaluate the impact on PFS of treatment strategy
* To estimate the Overall Survival (OS) in AYA with RMS
* To estimate the OS curve after relapse for patients who achieved complete remission during first line of treatment

Exploratory study Molecular profiling of RMS with the following subtypes: with fusiform cells (Embryonal RMS with fusiform cells vs adult RMS with fusiform cells or sclerosing) or pleomorphic (Embryonal RMS with anaplasia vs adult pleomorphic RMS) by RNAseq, and by CGH for ambiguous cases.

Methodology Clinical data from the different databases will be merged using a standardized format.

A pathology review of the slides is planned as well as a molecular characterization in borderline cases and unusual subtypes. MYOD1 mutations and molecular profile will be investigated for embryonal RMS.

Patient and treatment characteristics will be described with median, range, mean and standard deviation for continuous variables and in terms of frequency and percent of each modality for categorical variables.

PFS will be estimated using Kaplan-Meier method from diagnosis until relapse, progression or death from any cause. Patients alive without progression will be censored at the date of last news.

OS will be estimated using Kaplan-Meier method from diagnosis until death from any cause.

OS after relapse will be estimated using Kaplan-Meier method from the date of first relapse until the death whatever the cause. Patients alive will be censored at the date of last news.

Prognostic factors of PFS will be analyzed using Cox models after check of the proportional hazard assumption. The following factors will be evaluated:

* age: continuous or 15-18 vs 18-25
* tumor size: ≤ 5cm vs > 5cm
* primary tumor site according to the EPSSG classification: favorable (orbit, head and non parameningeal neck, paratesticular, vagina, uterus) vs unfavorable (head and parameningeal, vesico -prostatic, limb, other)
* IRS stage for primary tumor
* nodal and metastatic involvement at diagnostic
* histology (alveolar vs embryonic vs pleomorphic vs other)
* PAX3-FOXO1 and PAX7-FOXO1 fusion gene status, MYOD1 mutation The impact of treatment intervention on PFS will be evaluated using a Cox model stratified or adjusted over prognostic factors identified at the previous step.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 15 to 25 years old at diagnosis
* Patients registered in EpSSG RMS 2005 trial, or RRePS / NerSarc / Conticabase databases
* Over the period from 2006 to 2014
* Rhabdomyosarcoma histologically proven
* Localized or metastatic
* Histological review and molecular biology available
* No previous treatment except surgery
* No previous cancer
* Absence of known serious chronic illness
* Patient and/or parents information and non-opposition to data collection

Exclusion Criteria:

* Age over 25 years, or under 15 years
* Other histologies

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Patients aged from 15 to 25 years old at diagnosis
  * Patients registered in EpSSG RMS 2005 trial, or RRePS / NerSarc /
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years after diagnosis
  To estimate progression-free survival in AYA patients with RMS, according to clinical factors known as prognostic in children, and of biological factors (MYOD1 mutation in non-alveolar tumor; FOXO1).

SECONDARY OUTCOMES:
Clinical parameters of RMS in AYA | 9 months
  Clinical data from the different databases will be merged using a standardized format in order to describe the Clinical parameters of RMS in AYA
Biological parameters of RMS in AYA | 9 months
  Description of the RMS in AYA using biological characteristics (FOXO1, MYOD1 - where appropriate -, CGH-array profile)
therapeutic strategy | 9 months
  Description of the therapeutic strategy according to the different type of patients (paediatric, AYA, or adult):
Overall survival (OS) | 3 years after diagnosis
  OS will be defined as the time from diagnosis to death or last contact with the patient.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - BORDEAUX Bergonié, Bordeaux
  - Bordeaux Chu, Bordeaux
  - Brest Chu, Brest
  - LILLE Centre Oscar Lambret/ CHRU de Lille, Lille
  - LYON- Bérard, Lyon
  - MARSEILLE La Timone, Marseille
  - Montpellier Chu, Montpellier
  - MONTPELLIER ICM Val d'Aurelle, Montpellier
  - CHU de Nancy, Nancy
  - Nantes Chu, Nantes
  - NANTES Institut de Cancérologie de l'Ouest, Nantes
  - NICE CHU, Nice
  - NICE Centre Antoine Lacassagne, Nice
  - PARIS Curie, Paris
  - Poitiers Chu, Poitiers
  - Strasbourg Chru, Strasbourg
  - TOULOUSE Institut Claudius Regaud, Toulouse
  - TOURS CHU-Bretonneau/Hôp G de Clocheville, Tours
  - NANCY Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Villejuif Igr, Villejuif

REFERENCES:
- See also: Related Info — https://www.breastcancercare.org.uk/